CLINICAL TRIAL: NCT02963818
Title: Smartphone Technology Effects on Alcohol Drinking Among Young (STEADY) Adults Study
Brief Title: Smartphone Technology: Young Adult Drinking
Acronym: STEADY
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201600614-N; R21AA023368 (NIH)
Record Dates: First submitted 2016-11-08; First posted 2016-11-15 (Estimated); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Alcohol Use; Alcohol Drinking; Drinking Behavior
Keywords: Brief intervention; Harm reduction; Young adult; College Student
MeSH Terms: conditions — Alcohol Drinking; Drinking Behavior; Harm Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Smartphone breathalyzer device & app (Experimental): This is a small device that connects to a smartphone with an accompanying app that produces accurate breath alcohol readings when a user blows into a small tube attached to the device. Participants randomized to this study condition will have the opportunity to use this device and app during an alcohol drinking session in an actual bar and during a two-week field period.
  Interventions: Other: Smartphone breathalyzer device/app use
- BAC estimator app (Experimental): This is an app that produces estimated blood alcohol content (eBAC) readings based on sex, weight, number of drinks and time taken to consume drinks. Participants randomized to this study condition will have the opportunity to use this app during an alcohol drinking session in an actual bar and during a two-week field period.
  Interventions: Other: BAC estimator app use
- Text Messaging (Experimental): A procedure whereby one sends a text message to the phone one is using after each alcoholic drink. Participants randomized to this study condition will have the opportunity to the text messaging procedure during an alcohol drinking session in an actual bar and during a two-week field period.
  Interventions: Other: Text messaging procedure

INTERVENTIONS:
Other: Smartphone breathalyzer device/app use — Participants randomized to this condition will be able to blow into the smartphone breathalyzer after consuming each alcoholic drink, which produces an accurate breath alcohol reading on the app. These breath alcohol readings may inform participants' subsequent decisions regarding drinking.
  Arms: Smartphone breathalyzer device & app
Other: BAC estimator app use — Participants randomized to this condition will be able to make an entry into the BAC estimator app after consuming each alcoholic drink, which produces an estimated blood alcohol concentration based on the individual's sex, weight, number of alcoholic drinks and time spent drinking alcohol. These estimated blood alcohol concentrations may inform participants' subsequent decisions regarding drinking.
  Arms: BAC estimator app
Other: Text messaging procedure — Participants randomized to this condition will be instructed to send a text to a smartphone they will use for the study after each alcoholic drink. A consideration of the number of texts sent may inform participants' subsequent decisions regarding drinking.
  Arms: Text Messaging

SUMMARY:
Exploring technology based tools to reduce drinking is important. The purpose of this research study is to compare different BAC monitoring apps for their effects on alcohol drinking and ratings of usability among young adults.This study will be conducted in six phases: a web-based and in-person screening assessment; brief counseling session on the day before the alcohol drinking session; brief appointment on the day of the alcohol drinking session; alcohol drinking session; two-week field period; and a follow-up appointment. Participation in this study will last approximately two months.

ELIGIBILITY:
Inclusion Criteria:

* Be able to read/write English and complete study assessments
* Drink alcohol regularly

Exclusion Criteria:

* Test positive on a urine test for use of certain illegal drugs
* Undergraduate student enrolled at the University of Florida
* Graduate students from the College of Health and Human Performance at the University of Florida
* Pregnant, or currently breast feeding

Ages: 21 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2016-11; Primary Completion 2019-06-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Quantity of alcohol consumption | During one alcohol drinking session, an average of 2 hours
  Compare forms of mobile technology for their effects on alcohol consumption

SECONDARY OUTCOMES:
Quantity of alcohol consumption | two-week field period
  Compare forms of mobile technology for their effects on alcohol consumption

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Leeman, Ph.D., Principal Investigator — University of Florida
Locations (1):
- EDGE Laboratory, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leeman RF, Berey BL, Frohe T, Rowland BHP, Martens MP, Fucito LM, Stellefson M, Nixon SJ, O'Malley SS. A combined laboratory and field test of a smartphone breath alcohol device and blood alcohol concentration estimator to facilitate moderate drinking among young adults. Psychol Addict Behav. 2022 Sep;36(6):710-723. doi: 10.1037/adb0000780. Epub 2021 Nov 11. PMID 34766785